CLINICAL TRIAL: NCT02838732
Title: Investigation on the Effect of Carnitine Supplement on Gut Microbiota and TMAO Production Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201507055MINC
Record Dates: First submitted 2016-07-08; First posted 2016-07-20 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Dietary Exposure
Keywords: Gut microbiota; Trimethylamine N-oxide; L-carnitine supplementation; Oral carnitine challenge test

STUDY DESIGN:
Intervention Model Description: All participants received L-carnitine supplementation (500 mg per tablet per day, GNC) for one month. Oral carnitine challenge tests and fecal sampling were conducted both before and after the intervention.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-carnitine supplementation (Experimental): All participants received L-carnitine supplementation (500 mg per tablet per day, provided by GNC) for one month. Oral carnitine challenge tests and fecal sampling were conducted both before and after the intervention.
  Interventions: Dietary Supplement: L-carnitine supplementation (500 mg per tablet per day, purchased from GNC company)

INTERVENTIONS:
Dietary Supplement: L-carnitine supplementation (500 mg per tablet per day, purchased from GNC company)

SUMMARY:
In this project, the investigators aim to explore the impact of dietary L-carnitine supplementation on the TMAO production capacity of gut microbiota.

DETAILED DESCRIPTION:
Recent studies have established plasma trimethylamine N-oxide (TMAO) levels as a strong, independent risk factor for cardiovascular disease. TMAO is produced by the interaction between gut microflora and ingested L-carnitine from food. Research indicates that both plasma TMAO concentration and the TMAO production capacity of gut microbiota in vegetarians are significantly lower than in omnivores, likely due to the reduced L-carnitine intake in vegetarian diets. This study aims to explore the impact of L-carnitine supplementation on the TMAO production capacity of human gut microbiota and to identify TMAO-producing bacteria within the gut microflora. The study plans to recruit both omnivore and vegetarian volunteers to undergo a one-month L-carnitine supplementation, followed by an evaluation of changes in TMAO production using an oral L-carnitine challenge test, along with gut microbiota assessment. TMAO concentration will be measured using LC-MS/MS, and gut microbiome analysis will be conducted through shotgun metagenome sequencing. Bioinformatic analysis may reveal potential TMAO-producing bacteria. Understanding the changes in TMAO production and gut microbiota composition post-L-carnitine supplementation may enhance our knowledge of the interplay between L-carnitine supplements, TMAO, and gut microflora.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 20 to 65 years old
* no usage of antibiotics within one month
* no use of carnitine supplement within one month

Exclusion Criteria:

* having serious GI disorder
* medical history of myasthenia gravis
* history of diabetes,
* history of hyperparathyroidism,
* history of chronic kidney disease
* history of epilepsy
* history of severe anemia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-05-18; Primary Completion 2017-11-20 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
TMAO level | Before and 1 month after L-carnitine supplementation
  plasma and urine TMAO concentrations of oral carnitine challenge test
Compositional and functional alterations of gut microbiota | Before and 1 month after L-carnitine supplementation
  The compositional and functional changes of gut microbiota will be evaluated by shotgun metagenome sequencing. Taxonomy will be calculated as relative abundance of species-level genome bins (SGBs) and specific bacteria genes will be quantified as Reads Per Kilobase per Million (RPKM).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu WK, Chen CC, Liu PY, Panyod S, Liao BY, Chen PC, Kao HL, Kuo HC, Kuo CH, Chiu THT, Chen RA, Chuang HL, Huang YT, Zou HB, Hsu CC, Chang TY, Lin CL, Ho CT, Yu HT, Sheen LY, Wu MS. Identification of TMAO-producer phenotype and host-diet-gut dysbiosis by carnitine challenge test in human and germ-free mice. Gut. 2019 Aug;68(8):1439-1449. doi: 10.1136/gutjnl-2018-317155. Epub 2018 Oct 30. PMID 30377191